CLINICAL TRIAL: NCT04219436
Title: The Effect of Using Two Different Suturing Techniques on Free Gingival Marginal Stability After Esthetic Crown Lengthening for Treatment of Gummy Smile (Randomized Clinical Trial)
Brief Title: The Effect of Using Two Different Suturing Techniques on Free Gingival Marginal Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Hesham Mohamed, teaching assisatnt, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER16-35M
Record Dates: First submitted 2019-12-30; First posted 2020-01-07 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Altered Passive Eruption of Teeth
Keywords: esthetic crown lengthening; suturing technique; vertical mattress suturing technique; figure of eight suturing technique; tissue rebound; supracrestal gingival tissue; free gingival margin

STUDY DESIGN:
Intervention Model Description: 2 arms undergoing the same surgical procedure but with different suturing techniques for flap closure
Who Masked: Participant, Outcomes Assessor
Masking Description: The study consisted of two groups the number of patient was determined by sample size calculation through G power analysis (15 patients). Patients were randomly selected using computer generated randomization (www.randomizer.org).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vertical mattress suturing technique (Active Comparator): vertical mattress suturing technique is done to close the flap
  Interventions: Procedure: vertical mattress suturing technique
- figure of eight suturing technique (Active Comparator): figure of eight suturing technique is done to close the flap
  Interventions: Procedure: figure of eight suturing technique

INTERVENTIONS:
Procedure: vertical mattress suturing technique — vertical mattress suturing technique used for flap closure after esthetic crown lengthening
  Arms: vertical mattress suturing technique
Procedure: figure of eight suturing technique — figure of eight suturing technique used for flap closure after esthetic crown lengthening
  Arms: figure of eight suturing technique

SUMMARY:
Gummy smile is one of the major esthetic problems nowadays; it is due to several causes that either dental or skeletal. Etiology of the gummy smile is altered passive eruption, vertical maxillary excess, different gingival enlargement conditions, deficient maxillary lip length and excessive maxillary lip mobility, dento alveolar extrusion, combination of all these factors.

Altered passive eruption is considered to be one of the most major causes, it is classified into two types according to the location of the mucogingival junction with respect to the bone crest and each type has two subtypes . Esthetic crown lengthening is the treatment of choice for subtype B in both types as bone removal is mandatory to create a space for the biological width.

Most of the studies stated that there is some degree of relapse of the gingival tissues after the procedures in the follow ups, that relapse was related to the biotype of the gingival tissues, the flap placement close or far from the bone can be correlated to the suturing technique used for closure of the tissues.

In the investigator's study comparing of two different suturing technique was done to evaluated their effect on gingival tissue relapse, 30 patients (26 females and 4 males) were divided between 2 groups each group consisted of 15 patients. In the first group periosteal suturing technique was done in the second figure of eight (modified interrupted) suturing technique was.

Evaluation of the tissue relapse was done through the assessment of the amount of the attached gingival tissues level of gingival margin and marginal tissue contour before and after the surgery.

The results of the study showed that tissue relapse was more in the periosteal suturing technique group that was related to the pressure on the tissues due to the fixation of the suture at the periostium, the papillary tissue also showed more inflammation in the follow up period prior to suture removal. The figure of eight group showed less relapse and tissue inflammation as it prevents flap edge overlap and is tension free therefore better blood supply to the tissue.

Patients were generally satisfied post-surgical with their smile, gingival tissue visibility and teeth dimensions inspite of the relapse but it was better than prior to surgery. Also they would recommend it to other patients complaining from the same problem.

DETAILED DESCRIPTION:
Thirty patients (26 females, 4 males), who were candidates for esthetic crown lengthening, participated in this prospective clinical trial.

Group I (15 patients) (vertical mattress suturing technique) :

Esthetic crown lengthening procedure: internal bevel, sulcular and interdental incisions, flap elevation, bone removal then External vertical mattress suture was done (periosteal suture).

Group II (15 patients) (Figure of eight suturing technique) :

Esthetic crown lengthening procedure: internal bevel, sulcular and interdental incisions, flap elevation, bone removal then modified interrupted suture was done (Figure of eight suture).

ELIGIBILITY:
Inclusion Criteria:

* Patients complaining from gummy smile (altered passive eruption)
* Bone level is 2 mm or less from the cemento enamel junction
* Teeth included were free from any periodontal destruction
* Good compliance with the plaque control instructions following initial therapy.
* Availability for follow up and maintenance program

Exclusion Criteria:

* Presence of systemic diseases which could influence the outcome of the therapy (American society of anesthesiologists I, ASA I).
* Patient suffering from periodontitis stage 4 grade c.
* Presence of smoking habit.
* Presence of occlusion interference.
* Pregnant females and lactating females. .
* Vulnerable groups of patients (handicapped, mentally retarded, prisoners).
* Restored teeth.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
evaluation of the marginal soft tissue levels rebound | 6 months
  determination of soft tissue rebound: is measured as the difference between (the level of free gingival margin after suturing) and (the level of the free gingival margin 6 months post surgical) both measured from fixed reference point on the stent to the free gingival margin

SECONDARY OUTCOMES:
Supracrestal gingival tissue | 6 months
  the difference between the bone level and the free gingival margin (measured from a fixed reference point on the stent)
Patient satisfaction | at 6 months post surgical
  questionnaire (After surgery)
  * Is the patient satisfied with the gingival display during talking and smiling, teeth display during talking and smiling (not at all, slightly, somewhat, very and extremely).
  * How was the procedure experience (much worse, worse, same as I thought, better and much better).

CONTACTS AND LOCATIONS:
Overall Officials: ahmed gamal, professor, Study Director — faculty of dentistry ain shams university
Locations (1):
- Faculty of Dentistry Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
when the study is done the results will be published with the protocol
Supporting Information: Study Protocol, SAP
Time Frame: the data will be available starting next month and for 1 year
Access Criteria: the keywords esthetic crown lengthening, suturing techniques in dentistry

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT04219436/Prot_SAP_000.pdf